CLINICAL TRIAL: NCT02787681
Title: Multi-center Evaluation of the NEMO Gauge to Aid in Correct Positioning of the Endotracheal Tube After Intubation of Critically Ill Patients
Brief Title: Multi-center Evaluation of the NEMO Gauge to Aid in Correct Positioning of the Endotracheal Tube
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Loma Linda University (Other)
Responsible Party: Principal Investigator, H. Bryant Nguyen, Professor of Medicine, Loma Linda University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 5160137
Record Dates: First submitted 2016-05-23; First posted 2016-06-01 (Estimated); Results first posted 2020-11-09 (Actual); Last update posted 2020-11-09 (Actual); Status verified 2020-10

CONDITIONS: Respiratory Failure
MeSH Terms: conditions — Respiratory Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- NEMO Gauge (Experimental): Measurement and adjustment of endotracheal tube position by stylet.
  Interventions: Device: NEMO Gauge

INTERVENTIONS:
Device: NEMO Gauge — Measurement and adjustment of endotracheal tube position by stylet.

SUMMARY:
The aim of this study is to verify the safety and accuracy of an FDA-approved device called the NEMO™ Gauge to aide in the proper positioning of the endotracheal tube (ETT), inserted in the lungs of patients admitted to the intensive care unit. The hope is that the NEMO™ Gauge is able to properly determine the correct position of the endotracheal tube without the use of a chest radiograph (chest x-ray). The study investigators anticipate sixty-eight (68) subjects will participate in this study at three (3) study centers in the Inland Empire of Southern California, with subjects being enrolled at Loma Linda University Medical Center, Riverside University Medical Center and Loma Linda Veterans Affairs Hospital.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients ≥ 18 years of age admitted to the intensive care unit (ICU)
2. Patients who have been intubated or at high risk of being intubated, requiring confirmation of ETT position after intubation as determined by the clinical team
3. Endotracheal tube size 7.0 mm to 8.5 mm in diameter

Exclusion Criteria:

1. Patients with active hemoptysis
2. Patients with known tracheal or bronchial masses prior to endotracheal intubation
3. Patients with known tracheal or bronchial abnormalities requiring surgical repair

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2016-08-15 (Actual); Primary Completion 2017-07-14 (Actual); Study Completion 2017-07-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: H. Bryant Nguyen, MD, Principal Investigator — Loma Linda University
Locations (3):
- United States (3):
  - Loma Linda University Medical Center, Loma Linda, California
  - VA Loma Linda Healthcare System, Loma Linda, California
  - Riverside University Medical Center, Moreno Valley, California

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | NEMO Gauge
Started | 71
Completed | 69
Not Completed | 2

BASELINE CHARACTERISTICS:
Groups:
- NEMO Gauge: Baseline Characteristics
Arm/Group | NEMO Gauge
Number analyzed (Participants) | 69
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.2 (19.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22
  Male | 47
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
BMI [Mean (Standard Deviation); unit: kg/m2] | 31 (13.8)
Acute Respiratory Failure (Reason for Admission) [Count of Participants; unit: Participants] — Reason for Admission
  Participants | 52
Sepsis (Reason for Admission) [Count of Participants; unit: Participants] — Reason for Admission
  Participants | 14
Gastrointestinal (Reason for Admission) [Count of Participants; unit: Participants] — Reason for Admission
  Participants | 13
Neuromuscular (Reason for Admission) [Count of Participants; unit: Participants] — Reason for Admission
  Participants | 11
Shock on vasopressors (Reason for Admission) [Count of Participants; unit: Participants] — Reason for Admission
  Participants | 6
Cardiac (Reason for Admission) [Count of Participants; unit: Participants] — Reason for Admission
  Participants | 5
Renal (Reason for Admission) [Count of Participants; unit: Participants] — Reason for Admission
  Participants | 5
Other (Reason for Admission) [Count of Participants; unit: Participants] — Reason for Admission
  Participants | 2
Endotracheal Size 7 mm [Count of Participants; unit: Participants] | 2
Endotracheal Size 7.5 mm [Count of Participants; unit: Participants] | 41
Endotracheal Size 8 mm [Count of Participants; unit: Participants] | 26

OUTCOME MEASURES:

1. Primary Outcome: Number of Correct Endotracheal Tube Position
Description: The number of patients with correct Endotracheal tube position
Time Frame: Immediate, post-intervention
Measure: Count of Participants; unit: Participants
Arm/Group | NEMO Gauge
Number analyzed (Participants) | 69
Participants | 64

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | NEMO Gauge
All-Cause Mortality (participants affected / at risk) | 0/71
Serious Adverse Events (participants affected / at risk) | 0/71
Other Adverse Events (participants affected / at risk) | 0/71

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-07-21): https://cdn.clinicaltrials.gov/large-docs/81/NCT02787681/Prot_SAP_000.pdf